CLINICAL TRIAL: NCT04593290
Title: Listen Carefully: An Exploratory Study of the Association Between Listening Effort and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Denmark (Other)
Collaborators: Danish Dementia Research Centre (Network)
Responsible Party: Principal Investigator, Anja Maier, Professor, Deputy Head of Division, Group Leader, Technical University of Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19042404
Record Dates: First submitted 2020-06-05; First posted 2020-10-19 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Impairment, Mild; Hearing Loss
MeSH Terms: conditions — Cognitive Dysfunction; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild Cognitive Impairment (MCI) (Experimental): MCI is defined as an early stage of cognitive decline that lies between normal age-matched cognitive function and the onset of very mild forms of dementia, and is associated with a slight but noticeable decline in abilities such as memory and thinking skills. Listening effort testing (with pupillometry) and cognitive testing will be administered for this group - and after a 6-week period of hearing aid use, these measures will be re-tested.
  Interventions: Device: Oticon Opn S 1 miniRITE hearing aid
- Cognitively Healthy (Active Comparator): This group is 40-85 years old and has no significant neurological or psychiatric disease. Listening effort testing (with pupillometry) and cognitive testing will be administered for this group - and after a 6-week period of hearing aid use, these measures will be re-tested.
  Interventions: Device: Oticon Opn S 1 miniRITE hearing aid

INTERVENTIONS:
Device: Oticon Opn S 1 miniRITE hearing aid — Everyone who participates in Part 1 (listening effort testing and cognitive testing) will be invited to participate in Part 2 (hearing aids). It is not a requirement to participate in the administration, 6-week use, and re-testing procedures involved in Part 2 of the study. All cognitively healthy participants will be invited to participate, only MCI patients with a live-in informant will be given this opportunity. After ear measurement and dome and wire length selection, Oticon Opn S 1 miniRITE hearing aid fitting will occur wirelessly using Genie software, followed by hearing aid use instructions. The fitting will use Open domes, the standard NAL-NL2 protocol, and will increase gain seven steps on top of Real Ear Unaided Gain (REUG) from 750 Hz to 6 kHz.

SUMMARY:
This study aims to investigate the association between listening effort and cognitive function for both cognitively healthy individuals and for patients with Mild Cognitive Impairment (MCI) in mid-to-late stages of life, and furthermore to investigate listening effort and cognitive function after several weeks of hearing aid use. Listening effort is measured by the recording of peak pupil dilation during a sentence-final word identification and recall (SWIR) test, cognitive performance is measured using a battery of pen and paper cognitive tests, and hearing loss is measured with pure tone audiometry (PTA). A select number of participants in both the cognitively healthy and MCI group will be administered hearing aids, and the study will re-test both listening effort and cognitive performance.

DETAILED DESCRIPTION:
This is an exploratory proof-of-concept study and an exploratory intervention study with hearing aids in the context of listening effort. With a case (MCI) and control group (cognitively healthy), investigators will examine the associations between listening effort and cognitive function and assess the effect of hearing aid use on both listening effort and cognitive function test scores for those without hearing impairment. There is not sufficient literature to support a sample size calculation for this association study. Investigators will recruit approximately 50 participants. Half of these participants (n=25) will be individuals who have been diagnosed with MCI, according to the Winblad criteria (ICD10), with a Mini Mental State Examination (MMSE) score ≤ 26. The control group of participants (n=25) will be cognitively healthy individuals. All participants will undergo both listening effort testing, coupled with pupillometry and cognitive performance testing, based on a battery of pen-and-paper neuropsychological tests.

As investigators aim to measure cognitive effort exerted when listening and understanding speech in noise, is important that all study participants exhibit a normal sensitivity threshold within the ear canal. This will be assessed using Pure Tone Audiometry (PTA).

Assessment scores for cognitive function will be recorded in a clinical setting, and will be based on a battery of pen-and-paper neuropsychological cognitive tests. The Stroop Test, Trail Making Test (part A & B), Symbol Digit Modalities Test (SDMT), Verbal Fluency Tests (category: animals and lexical), Rey Complex Figure Test and Logical Memory Test (Part A) will be administered.

The objective measure of listening effort, pupil dilation, will be recorded as a measure of task performance accuracy and pupil dilation will be measured during a SWIR test, which is used to measure speech identification and recall in varying background noise. Prior to the SWIR test, participants undergo an adaptive Danish Hearing in Noise Test (HINT), comprising a list of equally intelligible sentences to be repeated in varying decibel (dB) levels of background noise to determine the individual's speech reception threshold (SRT) at 80% correct responses.

During the SWIR test, the participant is fitted with PupilLabs' eye-tracking system, an open source system consisting of clip-in eye tracking hardware to be placed in a Virtual Reality (VR) headset. To prevent floor and ceiling effects that are independent to baseline pupil size, the illumination within the VR display is individually adapted to the individual's midpoint prior to data collection between dim (~30 lux) and bright (~230 lux), with an average illuminance of 110 lux. A software suite allows the capture and post-processing of the data feed, including pupil diameter. For the purpose of this study, the PupilLabs software is controlled via a MATLAB interface.

Everyone who participates in Part 1 (listening effort testing and cognitive testing) will be invited to participate in Part 2 (hearing aids). It is not a requirement to participate in the administration, 6-week use, and re-testing procedures involved in Part 2 of the study. All cognitively healthy participants will be invited to participate, only MCI patients with a live-in informant will be given this opportunity. After ear measurement and dome and wire length selection, Oticon Opn S 1 miniRITE hearing aid fitting will occur wirelessly using Genie software, followed by hearing aid use instructions. The fitting will use Open domes, the second generation of the National Acoustic Laboratories (NAL) fitting protocol (NAL-NL2) and will increase gain seven steps on top of Real Ear Unaided Gain (REUG) from 750 Hz to 6 kHz.

ELIGIBILITY:
MCI group

Inclusion Criteria:

* Is 40-85 years old;
* Has no other significant neurological or psychiatric disease;
* Has normal hearing (0 - 25 dB thresholds from 250 -6 kHz) measured using PTA;
* Has normal or corrected to normal vision;
* Has an MCI diagnosis, according to Winblad criteria, with a score on the Mini Mental State Examination (MMSE) less than or equal to 26 (MMSE ≤ 26);
* Has a CDR = 0.5;
* Speaks Danish as native language
* (For part 2 of the study - hearing aid use) has a live-in informant.

Exclusion Criteria:

* Takes medication or treatment that could impact the pupillary dilation: eye drops (e.g. atropine or phenylephrine);
* Takes medication or treatment that could impact cognitive function;
* Abuses alcohol or drugs;
* Is unable to comply with study procedures.

Cognitively healthy group:

Inclusion criteria:

* Is 40-85 years old;
* Has a score above 26 on the Mini Mental State Examination (MMSE) (MMSE > 26);
* Has a CDR Global score = 0;
* Has no significant neurological or psychiatric disease;
* Has Normal hearing (0 - 25 dB thresholds from 250 -6 kHz) measured using PTA;
* Has Normal or corrected to normal vision;
* Speaks Danish as a native language.

Exclusion criteria:

* Meets the criteria for MCI (Winblad criteria) or dementia (ICD 10);
* Takes medication or treatment that could impact the pupillary dilation: eye drops (e.g. atropine or phenylephrine);
* Takes medication or treatment that could impact cognitive function;
* Abuses alcohol or drugs;
* Is unable to comply with study procedures.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Listening effort | Baseline, pre-intervention
  Listening effort will be measured by the percent of correctly recalled words in the SWIR test and the time-bound pattern in the pupil dilation traces during the SWIR test.
The Stroop Color and Word test | Baseline, pre-intervention
  Neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect.
  Measure: time (seconds) and number of mistakes.
  Increased time corresponds to poorer performance. Increased mistakes correspond to poorer performance.
Rey Complex Figure Test | Baseline, pre-intervention
  Neuropsychological assessment, administered by trained neuropsychologist, where examinees are asked to reproduce a complicated line drawing, first by copying it freehand and then drawing it from recall. This tests both recognition and recall, and uses visuospatial abilities, memory, attention, planning, working memory and executive functions.
  Measure: Accuracy scores between 0 and 2 on 18 figure elements (from 0 to a maximum of 36) on both copy and delayed recall
  Higher score = improved performance
Symbol-Digit Modalities Test | Baseline, pre-intervention
  Neuropsychological assessment commonly used in clinical and research settings to assess neurological dysfunction. The participant has 90 seconds to pair specific numbers with given geometric figures. Like other substitution tasks, performance is underpinned by attention, perceptual speed, motor speed, and visual scanning.
  Measure: Total score based on number of pairings made in 90 seconds ( maximum of 110 pairings).
  Higher score corresponds to improved performance.
Trail Making Test A and B | Baseline, pre-intervention
  Neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. Test A has participants follow numbers sequentially, while Test B has participants follow alternating numbers and letters, sequentially. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
  Measure: Test A - total time (seconds) required to connect 25 numbers, Test B - total time (seconds) required to connect 13 numbers and alphabet to letter H.
  Increased time corresponds to poorer performance.
Verbal Fluency Test (category and lexical) | Baseline, pre-intervention
  Participants are given 1 minute to produce as many unique words as possible within a semantic category (category fluency) or starting with a given letter (letter fluency). Category fluency tasks rely on language representations of semantic concepts, whereas lexical and action word task rely more on the central executive component of working memory.
  Measure: Number of unique words identified within 1 minute.
  More words correspond to improved performance.
Logical Memory Test A | Baseline, pre-intervention
  The Logical Memory test (part A) is a subtest of the Wechsler Memory Scale-Revised, and is a standardised assessment of narrative episodic memory. A short story is orally presented and the examinee is asked to recall the story verbatim. 25-35 minutes later, free recall of the story is again elicited (delayed recall), and a series of 30 questions are asked about the story.
  Measure: scores between 0 and 1 on specific pieces of the story (maximum score of 25) in both immediate and delayed recall. For the questions, a score of 0 or 1 is given to the corresponding 30 questions (maximum score of 30).
  Higher score corresponds to improved performance.

SECONDARY OUTCOMES:
Listening effort post-hearing aid use | Post-intervention, after 6 weeks of intervention (hearing aid use)
  Listening effort will be measured by the percent of correctly recalled words in the SWIR test and the time-bound pattern in the pupil dilation traces during the SWIR test.
Logical Memory Test A post-hearing aid use | Post-intervention, after 6 weeks of intervention (hearing aid use)
  The Logical Memory test (part A) is a subtest of the Wechsler Memory Scale-Revised, and is a standardised assessment of narrative episodic memory. A short story is orally presented and the examinee is asked to recall the story verbatim. 25-35 minutes later, free recall of the story is again elicited (delayed recall), and a series of 30 questions are asked about the story.
  Measure: scores between 0 and 1 on specific pieces of the story (maximum score of 25) in both immediate and delayed recall. For the questions, a score of 0 or 1 is given to the corresponding 30 questions (maximum score of 30).
  A higher score corresponds to improved performance
Verbal Fluency Test (category and lexical) post-hearing aid use | Post-intervention, after 6 weeks of intervention (hearing aid use)
  Participants are given 1 minute to produce as many unique words as possible within a semantic category (category fluency) or starting with a given letter (letter fluency). Category fluency tasks rely on language representations of semantic concepts, whereas lexical and action word task rely more on the central executive component of working memory.
  Measure: Number of unique words identified within 1 minute.
  More words corresponds to improved performance.
Trail Making Test A and B - post-hearing aid use | Post-intervention, after 6 weeks of intervention (hearing aid use)
  Neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. Test A has participants follow numbers sequentially, while Test B has participants follow alternating numbers and letters, sequentially. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
  Measure: Test A - total time (seconds) required to connect 25 numbers, Test B - total time (seconds) required to connect 13 numbers and alphabet to letter H.
  Increased time corresponds to poorer performance.
Symbol-Digit Modalities Test | Post-intervention, after 6 weeks of intervention (hearing aid use)
  Neuropsychological assessment commonly used in clinical and research settings to assess neurological dysfunction. The participant has 90 seconds to pair specific numbers with given geometric figures. Like other substitution tasks, performance is underpinned by attention, perceptual speed, motor speed and visual scanning.
  Measure: Total score based on number of pairings made in 90 seconds ( maximum of 110 pairings).
  Higher score corresponds to improved performance.
Rey Complex Figure Test | Post-intervention, after 6 weeks of intervention (hearing aid use)
  Neuropsychological assessment where participants are asked to reproduce a complicated line drawing, first by copying it freehand and then drawing it from recall. This tests both recognition and recall, and uses visuospatial abilities, memory, attention, planning, working memory and executive functions.
  Measure: Accuracy scores between 0 and 2 on 18 figure elements (from 0 to a maximum of 36) on both copy and delayed recall.
  Higher score corresponds to improved performance.
The Stroop Color and Word test | Post-intervention, after 6 weeks of intervention (hearing aid use)
  Neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect.
  Measure: time (seconds) and number of mistakes.
  Increased time corresponds to poorer performance. Increased mistakes correspond to poorer performance.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Maier, Ph.D., Principal Investigator — DTU - Technical University of Denmark
Locations (1):
- Copenhagen Memory Clinic, Rigshospitalet, Copenhagen, Region H, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pichora-Fuller MK, Kramer SE, Eckert MA, Edwards B, Hornsby BW, Humes LE, Lemke U, Lunner T, Matthen M, Mackersie CL, Naylor G, Phillips NA, Richter M, Rudner M, Sommers MS, Tremblay KL, Wingfield A. Hearing Impairment and Cognitive Energy: The Framework for Understanding Effortful Listening (FUEL). Ear Hear. 2016 Jul-Aug;37 Suppl 1:5S-27S. doi: 10.1097/AUD.0000000000000312. PMID 27355771
- [Background] Zekveld AA, Kramer SE, Festen JM. Cognitive load during speech perception in noise: the influence of age, hearing loss, and cognition on the pupil response. Ear Hear. 2011 Jul-Aug;32(4):498-510. doi: 10.1097/AUD.0b013e31820512bb. PMID 21233711
- [Background] Dawes P, Emsley R, Cruickshanks KJ, Moore DR, Fortnum H, Edmondson-Jones M, McCormack A, Munro KJ. Hearing loss and cognition: the role of hearing AIDS, social isolation and depression. PLoS One. 2015 Mar 11;10(3):e0119616. doi: 10.1371/journal.pone.0119616. eCollection 2015. PMID 25760329
- [Background] Panza F, Solfrizzi V, Logroscino G. Age-related hearing impairment-a risk factor and frailty marker for dementia and AD. Nat Rev Neurol. 2015 Mar;11(3):166-75. doi: 10.1038/nrneurol.2015.12. Epub 2015 Feb 17. PMID 25686757
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Griffiths TD, Lad M, Kumar S, Holmes E, McMurray B, Maguire EA, Billig AJ, Sedley W. How Can Hearing Loss Cause Dementia? Neuron. 2020 Nov 11;108(3):401-412. doi: 10.1016/j.neuron.2020.08.003. Epub 2020 Aug 31. PMID 32871106
- [Derived] Feldman A, Patou F, Baumann M, Stockmarr A, Waldemar G, Maier AM, Vogel A. Listen Carefully protocol: an exploratory case-control study of the association between listening effort and cognitive function. BMJ Open. 2022 Mar 9;12(3):e051109. doi: 10.1136/bmjopen-2021-051109. PMID 35264340